CLINICAL TRIAL: NCT00794638
Title: A Multicenter Phase I Clinical Trial to Assess the Safety of Two Consecutive Days of SyB L-0501 in Combination With Rituximab to Patients With Aggressive B-cell Non-Hodgkin's Lymphoma
Brief Title: A Phase I Clinical Trial of SyB L-0501 in Combination With Rituximab to Patients With Aggressive B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008002
Record Dates: First submitted 2008-11-18; First posted 2008-11-20 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Non-Hodgkin's Lymphoma; Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Diffuse Large B-Cell Lymphoma; Mantle cell Lymphoma; Transformed lymphoma, transformed to diffuse large B-cell lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SyB L-0501 — The administration of SyB L-0501 90 mg/m2 or 120 mg/m2/day on Day 2 and Day 3 will be followed by 18 days of observation. In the absence of adverse events or progressive disease, treatment will be repeated up to a maximum of 6 cycles, where 1 cycle is the 21-day treatment period (3 days of administration and 18 days of observation).
  Other Names: Bendamustine hydrochloride
Drug: Rituximab — The administration of rituximab 375 mg/m2 on Day 1 of each cycle will be followed by 18 days of observation. In the absence of adverse events or progressive disease, treatment will be repeated up to a maximum of 6 cycles, where 1 cycle is the 21-day treatment period (3 days of administration and 18 days of observation).

SUMMARY:
The purpose of this study is to assess the safety of SyB L-0501 in combination with Rituximab to patients with aggressive B-cell non-Hodgkin's lymphoma, and to explore the recommended dose for the Phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Aggressive B-cell non-Hodgkin's lymphoma patients with prior therapy who satisfy the conditions listed below. No restrictions regarding gender.

* Patients with the following histologically confirmed CD20(+) B-cell non-Hodgkin's lymphoma:

  1. Diffuse large B-cell lymphoma
  2. Mantle cell lymphoma
  3. Transformed lymphoma
  4. Follicular lymphoma (Grade 3)
* Fail to CR in prior chemotherapy, or relapse following CR or recurrence following PR.
* Patients who are judged to carry no effect from the prior therapy (cancer chemotherapy, antibody therapy and radiation/ radiotherapy.
* Patients aged from 20 to 75 years at the time informed consent is obtained
* Patients with adequately maintained organ functions (e.g., bone marrow, heart, lung, liver, and kidney functions)
* Patients who can be hospitalized during the first cycle
* Patients capable of personally giving voluntary informed consent in writing to participate in the study

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded.

* Patients with serious complications (hepatic or renal failure)
* Patients with complications or medical history of serious cardiac disease (e.g., myocardial infarction, ischemic heart disease)
* Patients with serious gastrointestinal symptoms (e.g., severe nausea, vomiting, or diarrhea)
* Patients positive for HBs antigen, HCV antibody, or HIV antibody
* Patients who received other investigational drug or unapproved medication within 3 months before registration in this study
* Patients who had history of hematopoietic stem cell transplantation or radioimmunotherapy
* Patients who are pregnant, of childbearing potential, or lactating
* Patients, whether male or female, who do not agree to contraception
* Patients otherwise judged by investigator or sub investigator to be unsuitable

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Treatment period

SECONDARY OUTCOMES:
CR rate and the overall response rate, determination by Independent Review Committee | Treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Kensei Tobinai, MD, Ph D, Study Chair — National Cancer Center Hospital
Locations (4):
- Japan (4):
  - Nagoya, Aichi-ken
  - Isehara, Kanagawa
  - Kyoto, Kyoto
  - Chuo-ku, Tokyo